CLINICAL TRIAL: NCT02244307
Title: Evolution of Patients Suffering From Benign Prostatic Hyperplasia (BPH) Treated With Alpha-adrenergic Blockade (JOSEPHINE)
Brief Title: Observational Study in Patients Suffering From Benign Prostatic Hyperplasia Treated With Alpha-adrenergic Blockade
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.28
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Adrenergic alpha-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with BPH treated with alpha-andrenergic blockade
  Interventions: Drug: alpha-adrenergic blocker

INTERVENTIONS:
Drug: alpha-adrenergic blocker

SUMMARY:
The primary objective of this observational study was the assessment of prognosis factors for having recourse to prostatic surgery in patients with BPH who were administered class-1 alpha blockers. The secondary objectives were the assessment of the time from alpha-adrenergic blockade treatment initiation to surgery and the evolution of patients during the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with BPH for whom alpha-blocker treatment is indicated
* Patients who are already on class-1 alpha-blockers can only participate in the study if all information required is known and/or available

Exclusion Criteria:

* Patient's follow-up not possible
* Patients participating in another study
* History of BPH surgery
* Prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with BPH for whom alpha-blockade treatement is indicated recruited at general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 4561 (Actual)
Dates: Start 2000-01; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Assessment of prognosis factors for having recourse to prostatic surgery | up to 2 years

SECONDARY OUTCOMES:
Time form alpha-adrenergic blockade treatment initiation to surgery | up to 2 years
Occurrence of concomitant BPH diseases | up to 2 years
Total International Prostate Symptom Score (IPSS) | up to 2 years
Percentage of patients with ongoing BPH treatment | up to 2 years